CLINICAL TRIAL: NCT02120430
Title: Promoting Effective Child Development Practices in the First Year of Life Through a Video Administered at Two Different Times. A Randomized Controlled Trial
Brief Title: Promoting Child Development Practices in the First Year of Life Through a Video Administered at Two Different Times
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RC 60/07
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Early childhood; Audiovisual materials; Parent-child interaction; Parenting programs; Timing
MeSH Terms: conditions — Behavior | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early administration of the video (Active Comparator): Video delivered at one month of child's life
  Interventions: Other: Video
- Late administration of the video (Experimental): Video delivered at seven months of child's life
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — The video was developed by a multidisciplinary team (psychologists, paediatricians, filmmaker). It was conceived as an aid to parenting in the first year of life, providing opportunities for parents to look at their own experiences. The video lasts 24 minutes and describes "the birth of a new relationship" between primary caregivers and their babies, in chronological order, starting from late pregnancy to the end of the first year. Caregiver-child interactions are shown from early contact after delivery to common care practices, with an emphasis on four specific activities, which are believed to improve child development and caregiver-child interaction: reading aloud to the baby, exposure to songs, rhymes and music, promotion of early socialization for parents and for children.

SUMMARY:
There is an increasing need for parenting programs aimed at promoting parent-child interaction. A variety of interventions have been proposed. The use of audiovisual materials for parents has been shown to be effective but limited information is available on the optimal timing for its use, particularly for new parents during the first year of life of their children.

Based on the hypothesis that the effectiveness of information provided to first-time parents in modifying their knowledge, attitudes and intentions regarding rearing practices may depend on when the information is delivered, we designed an open randomized controlled trial to compare the effectiveness of administering a video at two different times, i.e. at one and seven months of age of the child.

The video addressed four specific activities related to early child development: reading aloud to the baby, early exposure to music, promotion of early socialization for parents and for children.

ELIGIBILITY:
Inclusion Criteria:

* first parenting experience
* local residence
* no major health or psychosocial problems in parents and in the newborn
* no delay in discharge from the maternity ward
* adequate knowledge of Italian

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Parental knowledge, attitudes and intentions | 15 days after being exposed to the intervention
  Closed-ended questions about the four specific activities examined (reading aloud, exposure to music, caregiver and child early socialization) collected through a researcher-administered structured questionnaire

SECONDARY OUTCOMES:
Feelings elicited | 15 days after being exposed to the intervention
  Closed-ended questions collected through a researcher-administered structured questionnaire. Eight categories of emotions were evaluated: happiness, sadness, fear, rage, guilt, sense of competence, lack of self-confidence, and sense of inadequacy

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Tamburlini, MD, PhD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

REFERENCES:
- [Derived] Roia A, Paviotti E, Ferluga V, Montico M, Monasta L, Ronfani L, Tamburlini G. Promoting effective child development practices in the first year of life: does timing make a difference? BMC Pediatr. 2014 Sep 5;14:222. doi: 10.1186/1471-2431-14-222. PMID 25193490